CLINICAL TRIAL: NCT05893251
Title: Effectiveness of Cervical Treatment in Wind Musicians With Temporomandibular Dysfunction
Acronym: ANAISATM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANAISATM; ANAISATM (Other: UNIVERSITY OF MURCIA)
Record Dates: First submitted 2023-05-29; First posted 2023-06-07 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2018-03

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
Keywords: TEMPOROMANDIBULAR JOINT; Cervical Posture; wind Musician
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: The present study is an experimental, analytical, longitudinal, and prospective controlled randomized clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Using the "Random Team Generator" mobile application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocol group (Active Comparator): The treatment plan includes active postural exercises for the cervical spine.
  Interventions: Other: Postural exercises
- Manual therapy group (Experimental): The treatment plan includes active postural exercises and manual therapy for the cervical spine.
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Manual therapy — Within the manual therapy protocol carried out in the experimental group, we performed a series of passive maneuvers. The patient remains in supine position on a treatment table throughout the treatment, while the therapist sits at the head of the patient on a stool. The sequence of application is as follows:
  Suboccipital inhibition technique Cervical spinal mobilization Posterior fascia stretching
  Arms: Manual therapy group
Other: Postural exercises — The treatment plan includes active postural exercises for the cervical spine.
  Arms: Protocol group

SUMMARY:
Temporomandibular dysfunction (TMD) consists of a series of multifactorial signs and symptoms that occur in the orofacial region, with pain being the most common symptom. There is a close biomechanical and anatomical relationship between the cervical region and the temporomandibular joint (TMJ) through the trigemino-spinal nucleus.

Objectives: To comparatively assess the improvement in subjects with TMD when adding cervical manual therapy to a postural treatment. Additionally, to determine if both cervical treatments separately produce changes in the TMJ.

Materials and methods: An experimental study of randomized controlled clinical trial type was conducted. The study involved 30 wind instrument players randomly assigned to an experimental group (EG) and a control group (CG). After obtaining consent, measurements were taken for maximum mouth opening (MMO), cervical range of motion, and pain threshold to pressure (PTP) in the masseter and temporalis muscles. Both groups underwent active cervical postural treatment for 4 weeks, and the EG additionally received a cervical manual therapy protocol. An initial assessment was conducted before the intervention, and a final assessment was done one week after the last intervention. The statistical program SPSS was used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance of written informed consent.
* Playing a wind instrument.
* Age between 18-40 years.
* Pain in the cranio-cervico-mandibular region and/or masticatory muscles.
* Hypertrophy in the masticatory muscles.

Exclusion Criteria:

* History of trauma and/or fracture in the cranial and/or facial region.
* Rheumatic injury or degenerative disease.
* Surgical intervention on the temporomandibular joint (TMJ).
* Malformations of the cervical or cranial spine.
* Vestibular, circulatory, or neurological disorders.
* Degenerative or infectious joint diseases.
* Current orthodontic treatment.
* Receiving physiotherapy treatment during the two weeks prior to the study or during the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Cranio facial pain and disability inventory | a week after treatment
  CF-PDI (Craniofacial Pain and Disability Inventory): This questionnaire focuses on pain as a common symptom of TMD (Temporomandibular Disorders). It is self-administered and designed to assess patients' perception of their physical and psychosocial health in relation to craniofacial pain. It consists of 21 questions regarding the impact of pain on activities involving the use of the temporomandibular joint, with a scoring range from 0 to 63 in ascending order, where 0 indicates no impact and 63 indicates maximum impact. This questionnaire demonstrates good structure, internal consistency, reproducibility, and validity, making it an objective tool that can be used in research and clinical practice for evaluating patients with craniofacial pain and disability. It is easy to administer and requires a short amount of time. The CF-PDI was created and developed in Spain, based on a biopsychosocial approach.

SECONDARY OUTCOMES:
Maximum mouth opening. | a week after treatment
  The measurement of maximum mouth opening (MMO) is the distance in centimeters between the upper and lower incisor teeth when the subject actively opens their mouth.

OTHER OUTCOMES:
Pain pressure threshold in myofascial trigger points of the masticatory muscles. | a week after treatment
  In TMD, myofascial pain of the masticatory muscles is the most relevant clinical entity that affects the masticatory system. It will be measured using a pressure algometer.

CONTACTS AND LOCATIONS:
Locations (1):
- University Of Murcia, Murcia, Spain